CLINICAL TRIAL: NCT06830811
Title: Precision Assessment of Bone Mineral Density (BMD) Measurement With EOSedge™ - BMD Precision Study
Brief Title: Bone Mineral Density Precision Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alphatec Spine, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ATEC.EOS-2403
Record Dates: First submitted 2025-02-12; First posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Indicated for EOSedge Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Subjects indicated for EOSedge imaging (Other): Subject receiving EOSedge imaging as SOC will also receive an additional EOSedge scan.
  Interventions: Radiation: EOSedge imaging

INTERVENTIONS:
Radiation: EOSedge imaging — Full body or full spine image

SUMMARY:
The purpose of this research is to collect medical imaging data to allow for the comparison of bone mineral density measurements from two low-dose x-ray exams. The main question it aims to answer is:

What is the precision measurement between the BMD assessments from 2 x-ray exams?

DETAILED DESCRIPTION:
This is a single-center, prospective, precision study of 30 subjects indicated for radiography using EOSedge biplanar full-body or full-spine imaging.

From the potential pool of EOSedge examinees, screening data will be reviewed to determine further eligibility. Subjects who sign an informed consent form and meet all inclusion criteria and none of the exclusion criteria will be asked to participate in the study.

Subjects who consent to participate will be enrolled from the time of consent through completion of evaluable image acquisition which will include both EOSedge exams.

EOSedge exams will be performed as is typical for the evaluation of spinal and/or other orthopaedic conditions, and the output will be collected for post-hoc computation of BMD.

The second EOS exam will be study prescribed and performed immediately after the first exam, with the operator repositioning the subject between acquisitions, i.e., removing the subject from the scanner and repositioning between exams.

In addition to the radiographic imaging from which spinal/postural alignment parameters may be obtained, some demographic and diagnostic details about the subject will be captured via study-specific case report forms (CRFs). Subjects will also complete a questionnaire that every subject fills out prior to having a bone mineral density scan according to ISCD guidance.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects indicated for full-spine or whole-body radiography via EOSedge 2E biplanar imaging (e.g., in the preoperative evaluation of spine and/or other orthopaedic conditions)
2. Male or female subjects who are at least 20 years of age at the time of imaging acquisition
3. Written informed consent obtained from the potential subject or the subject's legal representative and ability for the subject to comply with the requirements of the study

Exclusion Criteria:

1. Subjects who have been administered contrast agents or radionuclides within 7 days prior to scheduled radiographic imaging (EOS and DXA)
2. Subjects who are pregnant or wanting to become pregnant during the timeframe of study participation (due to risks associated with radiographic imaging)
3. Subjects with a BMI ≥ 35 kg/m2
4. Subjects known to have severe degenerative changes or fracture deformity in the measurement area (i.e., lumbar spine L1-L4, bilateral femoral neck/trochanter; note that unilateral femoral evaluation is acceptable), as defined by the Investigator's determination of the likelihood of reasonably assessing bone mineral density of those areas
5. Subjects known to have implants, hardware, devices, or other foreign material in the measurement area (i.e., lumbar spine L1-L4, bilateral femoral neck/trochanter; note that unilateral femoral evaluation is acceptable)
6. Subjects unable to attain correct position and/or remain motionless for the measurement (e.g., subjects unable to stand unassisted in the EOS unit, or to lie appropriately in the DXA scanner)
7. Subjects known to have extra or missing lumbar vertebrae (i.e., more or fewer than 5 mobile lumbar segments)
8. Subjects participating in another clinical study which may compromise this study's results or compliance with this study's procedures
9. Subjects with presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the subject or the quality of the data

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-13 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
AP Spine BMD Precision | 1 day
  Calculation of EOSedge BMD from the 2 exams will be post-processed from the bi-planar EOSedge 2E radiographs, and is measured in g/cm² surface mass on four lumbar vertebrae (L1-L4) in the anteroposterior (AP) projection. Precision error will be calculated from the 2 exams.

SECONDARY OUTCOMES:
Hip BMD Precision | 1 day
  Calculation of EOSedge BMD from the 2 exams will be post-processed from the bi-planar EOSedge 2E radiographs, and is measured in g/cm² surface mass at the hip (femoral necks). Precision error will be calculated from the 2 exams.
Lateral L2-L3 Precision | 1 day
  Calculation of EOSedge BMD from the 2 exams will be post-processed from the bi-planar EOSedge 2E radiographs, and is measured in g/cm² surface mass at the spine (lateral L2-L3). Precision error will be calculated from the 2 exams.

CONTACTS AND LOCATIONS:
Locations (1):
- OrthoIndy, Fishers, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided